CLINICAL TRIAL: NCT01565538
Title: A Randomized Phase II Trial of Erlotinib Versus Pemetrexed as Second-Line Therapy in Treating Patients With Advanced EGFR Wild-Type and EGFR FISH-Positive Lung Adenocarcinoma
Brief Title: Erlotinib Versus Pemetrexed as Second-Line Therapy in Treating Patients With Advanced Lung Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Si-Yu Wang (Other)
Responsible Party: Sponsor-Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: wsy001
Record Dates: First submitted 2012-03-22; First posted 2012-03-28 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Lung Cancer
Keywords: Cancer; Non-small-cell lung cancer; Adenocarcinoma; EGFR gene mutation; Chemotherapy; Pemetrexed; Erlotinib
MeSH Terms: conditions — Lung Neoplasms; Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma | interventions — Erlotinib Hydrochloride; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erlotinib (Experimental): Erlotinib at the dose of 150 mg orally once a day continually until progression.
  Interventions: Drug: Erlotinib
- Pemetrexed (Experimental): Pemetrexed at the dose of 500mg/m2 IV infusion every 3 weeks until progression.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Erlotinib — 150 mg Given orally
  Other Names: Tarceva
  Arms: Erlotinib
Drug: Pemetrexed — 500mg/m2 Given IV
  Other Names: ALIMTA
  Arms: Pemetrexed

SUMMARY:
Both pemetrexed and erlotinib are second-line treatment options for patients with advanced non-small cell lung cancer. It is controversial that whether it is necessary to detect epidermal growth factor receptor (EGFR) mutation status for the EGFR-targeted therapy after the failure of standard chemotherapy. The role of EGFR gene copy number as a predictive marker remains controversial. Therefore, we investigate the efficacy of erlotinib and pemetrexed as second-line therapy in treating in patients with EGFR wild-type and EGFR FISH-positive advanced lung adenocarcinoma.

DETAILED DESCRIPTION:
Standard first-line treatment for advanced-stage non-small cell lung cancer (NSCLC) usually consists of platinum-based doublet chemotherapy, but progression ultimately occurs for most patients. Second-line treatment options available to patients who suffer failure of first-line treatment include further chemotherapy (docetaxel and pemetrexed) or targeted therapy. Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) show great efficacy in patients with advanced NSCLC with EGFR mutation. High EGFR gene copy number was associated with great sensitivity and prolonged progression-free survival of NSCLC from EGFR-TKIs. This phase II study was designed to assess the efficacy and safety of erlotinib compared with pemetrexed as second-line treatment for EGFR wild-type and EGFR FISH-positive lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Lung adenocarcinoma
* Wld-type EGFR
* Stage IIIB/IV
* Failure to prior chemotherapy
* Life expectancy of more than 3 months
* Tissue sample desired for genomic study
* Age ≥ 18 years
* Performance status (WHO) < 3
* Adequate bone marrow function (absolute neutrophil count > 1000/mm^3, platelet count > 100000/mm^3, hemoglobin > 9gr/mm^3)
* Adequate liver (bilirubin < 1.5 times upper limit of normal and SGOT/SGPT < 2 times upper limit of normal) and renal function (creatinine < 2mg/dl)
* Presence of two-dimensional measurable disease. The measurable disease should not have been irradiated
* Informed consent

Exclusion Criteria:

* Have previously received pemetrexed or TKIs
* Other concurrent uncontrolled illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-12; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Si-Yu Wang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li N, Ou W, Yang H, Liu QW, Zhang SL, Wang BX, Wang SY. A randomized phase 2 trial of erlotinib versus pemetrexed as second-line therapy in the treatment of patients with advanced EGFR wild-type and EGFR FISH-positive lung adenocarcinoma. Cancer. 2014 May 1;120(9):1379-86. doi: 10.1002/cncr.28591. Epub 2014 Jan 30. PMID 24481719

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib | Pemetrexed
Started | 61 | 62
Completed | 61 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Pemetrexed | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Continuous [Median (Full Range); unit: years] | 54.3 [30 to 74] | 55.1 [33 to 75] | 54.7 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 40 | 39 | 79
ECOG PS [Number; unit: participants] — Eastern Cooperative Oncology Group performance status. ECOG 0=Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours.
  participants
    0,1 | 57 | 59 | 116
    2 | 4 | 3 | 7
Smoking status [Number; unit: participants]
  Never | 15 | 17 | 32
  Former | 7 | 5 | 12
  Current | 39 | 40 | 79
Stage [Number; unit: participants] — Tumors were classified according to the 1997 International System for Staging Lung Cancer. Reference: Mountain CF. Revisions in the International System for Staging Lung Cancer.Chest.1997;111:1710-1717.
  participants
    IIIB | 4 | 6 | 10
    IV | 40 | 38 | 78
    Recurrent | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the date of randomization to the date of tumour progression or death from any cause, assessed until at least 12 months after randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Pemetrexed
Number analyzed (Participants) | 61 | 62
months | 4.1 [1.6 to 6.6] | 3.9 [2.7 to 5.1]

2. Secondary Outcome: Best Tumor Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From the date of randomization, assessed every 6 weeks, until at least 12 months after randomization.
Measure: Number; unit: participants
Arm/Group | Erlotinib | Pemetrexed
Number analyzed (Participants) | 61 | 62
participants
  Objective response | 12 | 5
  No objective response | 49 | 57

3. Secondary Outcome: Overall Survival
Time Frame: From date of randomization until the date of death from any cause, assessed until at least 12 months after randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Pemetrexed
Number analyzed (Participants) | 61 | 62
months | 11.7 [7.5 to 15.9] | 13.4 [9.2 to 17.7]

ADVERSE EVENTS:
Arm/Group | Erlotinib | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/62
Other Adverse Events (participants affected / at risk) | 45/61 | 43/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=61) | Pemetrexed (N=62)
Rash (Skin and subcutaneous tissue disorders) | 33 | 4
Diarrhea (Gastrointestinal disorders) | 10 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Anorexia (Gastrointestinal disorders) | 6 | 9
Nausea (Gastrointestinal disorders) | 1 | 15
Constipation (Gastrointestinal disorders) | 0 | 4
Fatigue (General disorders) | 12 | 16
Infection (Infections and infestations) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 4 | 3
Headache (Nervous system disorders) | 1 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Paronychia (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes